CLINICAL TRIAL: NCT02425488
Title: Nursing Therapeutics Education and Heart Failure (HF): an Experimental Study
Brief Title: Nursing Therapeutics Education and Heart Failure (HF): a Study Protocol
Acronym: NEHF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasability phase completed: Cost Evaluation
Sponsor: University of Turin, Italy (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Prof. Maria Michela Gianino, Professor in Hygiene and Public Health, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HFICD
Record Dates: First submitted 2015-04-20; First posted 2015-04-24 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Heart Failure; Arrhythmia
Keywords: Nursing; Outcome and Process Assessment; Cardiac Resynchronization Therapy Devices; Heart Failure; Education
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nursing therapeutics education (Experimental): People who are educated by the nurse (Behavioral intervention: Nursing therapeutics education) and follow all the program (12 months)
  Interventions: Behavioral: Nursing therapeutics education
- Non NET (No Intervention): People who receive basic information without follow the educational program but clinically controlled

INTERVENTIONS:
Behavioral: Nursing therapeutics education — Educational intervention will focus on
  1. Appropriate lifestyles
  2. Early recognition of signs/prodromal symptoms of HF
  3. Early recognition of signs of inflammation of the ICD-pocket
  4. Good management of the device
  1) Therapy, body weight, diet, smoking, alcohol, rest, exercise, job and sex 2) Dyspnea, edema and fovea, rapid weight gain, loss of appetite, fatigue, asthenia, insomnia, mental confusion 3) Signs and symptoms of inflammation: hyperpyrexia, rubor, dolor, calor and tumor 4) Identification tag, vibration, metal detectors, air travel, use of electronic devices, diagnostic PET and MRI
  Arms: Nursing therapeutics education

SUMMARY:
Purpose: Heart Failure (HF) is a clinical multifactorial syndrome, it can cause arrhythmias for which international guidelines suggest the implantation of an implantable cardiac defibrillator (ICD). The educational nursing program would improve clinical outcomes in patients with HF and ICD like control their sickness, known and acknowledge symptoms, improve their skills to self-care.

The main aim of this study is to assess how much the nursing-therapeutics skills and an educational intervention, in patients with HF during the follow-up period after the implantation of ICD reduces clinical costs, re-hospitalizations, and mortality at 180 days.

Methods: The investigators start a multicenter randomized clinical trial. The sample is made of 128 subjects (64 patients treatment group and 64 control group). The investigators measured the self-care level administering to HF patients the "Self-Care of Heart Failure Index (SCHFI) v. 6.2", and the self-perception of own life quality using a Numeric Rating Scale from 0 to 100. Secondary outcomes recorded are i) the numbers of accesses to the ED (Emergency Department) and/or hospitalizations during the follow-up period, ii) mortality rate due to HF, and iii) infection rate of the device pocket.

Data Analysis: Categorical variables will be presented in terms of frequencies and percentages. The statistical power was fixed at the 80%. Data will be considered significant for a p-value ≤ 0.05. The Cox proportional hazards model will be used to analyze mortality in subjects involved in the educational program.

DETAILED DESCRIPTION:
Aims of the study The aim of this study is to examine the effects of a nursing intervention consisting of sanitary-therapeutic education during the follow-up period after the implantation of a defibrillator (ICD) in patients with congestive heart failure.

The effectiveness of the educational intervention will be assessed on the basis of the level of "self-care" in every individual and their lifestyle as well as on mortality rates, readmission to the hospital and ICD pocket infection.

Educational intervention will focus on

1. Appropriate lifestyles
2. Early recognition of signs/prodromal symptoms of HF
3. Early recognition of signs of inflammation of the ICD-pocket
4. Good management of the device

<!-- -->

1. Therapy, body weight, diet, smoking, alcohol, rest, exercise, job, and sex
2. Dyspnea, edema, and fovea, rapid weight gain, loss of appetite, fatigue, asthenia, insomnia, mental confusion
3. Signs and symptoms of inflammation: hyperpyrexia, rubor, dolor, calor and tumor
4. Identification tag, vibration, metal detectors, air travel, use of electronic devices, diagnostic PET and MRI

   Materials and methods A multicenter randomized controlled study will be performed. The research project will involve two clinical centers in northern Italy: the "Città della Salute e della Scienza" University Hospital of Turin, which includes the "Molinette" Hospital (coordinator center), and the TO3 ASL, which includes the "Associated Hospitals of Rivoli".

   Subject recruitment and data collection will take place until data saturation is achieved, with an estimated period of approximately 12 months from the beginning of the study.

   Participants

   Inclusion criteria:
   * Patients affected by heart failure following elective hospitalization during which an ICD was implanted on an arrhythmic and/or ischemic basis.
   * Patients who have given written consent for the research.

   Exclusion criteria:
   * Patients with syndromes and diseases that compromise their understanding of information, learning and all cognitive activities in general.
   * Minors.

   Primary outcome measures • Self-care levels (measured using the Self-Care Heart Failure Index, SCHFI v 6.2)

   • Quality of life perception (measured using a numerical rating scale from 0 to 100)

   Secondary outcome measures • Number of visits to the ED (Emergency Department) and/or hospitalizations during the follow-up period after the implantation of a defibrillator (ICD).

   • Mortality rate at 180 days after the implantation of the ICD due to HF-related causes.

   • Infection rate in the device pocket.

   Data, sources and collection tools • Socio-demographic and clinical data: For all of the included patients, demographic (gender, age, educational level, marital status, country of birth (Italian citizens or foreigners), social (through a family context survey) and clinical (classification of HF using the NYHA classification, the implantation date and type of ICD, the execution of and the changes in laboratory tests and electrocardiograms results, number of perceived discharges) data will be recorded. Data on the patient's diagnosis and possible associated diseases will be obtained through the analysis of clinical documentation and will be record in accordance with the International Statistical Classification of Diseases and Related Health Problems, 9th Revision (ICD-IX).

   • Economic data: For patients included in the study, the following data will be collected:

   • economic activity, occupational qualifications (if employed/ex-employed);
   * visits to the ED and/or hospitalizations during the follow-up period, verified through analysis of administrative documentation certifying visits and admissions (Verbal First Aid and Medical record);
   * the presence of a companion for the patients during their stay in the ED or hospital as well as their economic activity and professional qualifications;
   * any costs directly incurred by the patient or companion;
   * time spent by the nursing figure in providing therapeutic education. From society's point of view, the benefits received in the ED and hospitalizations will be assessed according to the charge currently in force in Italy. Indirect costs, represented by the time spent by the patient, and costs related to the time spent by caregivers will be valorized using values published by official sources such as ISTAT. Costs directly charged to the patient will be valued on the basis of the stated cost. Finally, the cost of time spent in educational activities will be assessed using the hourly average cost of a nurse and/or doctor in the clinical centers that participate in this study.
   * Self-Care Heart Failure Index (SCHFI) version 6.2. A tool validated in the Italian context that allows evaluation of a patient's awareness and capacity for self-care11. The obtained responses are organized on a four-level Likert scale (1 = never, 4 = every day). Specifically, this instrument is divided into three sections:

   Section A: (questions 1 to 10) investigates self-care skills; Section B: (questions 11 to 16) investigates an individual's symptomatology recognition skills; Section C: (questions 17 to 22) investigates the self-confidence related to self-care skills in detail.

   The total score is computed in the following manner:

   Section A: 10 is subtracted from the sum of the section results considering answers 1 to 10, and the result is multiplied by a coefficient of 3.33; Section B: 4 is subtracted from sum of the section results considering answers 11 to 16, and the result is multiplied by a coefficient of 5; Section C: 6 is subtracted from sum of the section results considering answers 17 to 22, and the result is multiplied by a coefficient of 5.56 All of the results have to be considered in terms of percentages. If the percentages for individual sections are all higher than the cut-off value (70%), then according to the literature11, the level of self-care is considered adequate. Otherwise, for lower values, the section showing an insufficient result will be strengthened.
   * Numeric Rating Scale: scale from 0 to 100 used for subjective measurement of the perceived quality of life. This tool will be evaluated by a committee of experts using a pre-test, which is currently under way.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by heart failure following elective hospitalization during which an ICD was implanted on an arrhythmic and/or ischemic basis.
* Patients who have given written consent for the research.

Exclusion Criteria:

* Patients with syndromes and diseases that compromise their understanding of information, learning and all cognitive activities in general.
* Minors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2017-10-29 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Self-care levels (Self-Care Heart Failure Index (SCHFI) version 6.2) | 12 months
  Increase of the Self Care competence, management and confidence with heart failure and the cardiac device

SECONDARY OUTCOMES:
Quality life perception | 12 months
  Increase in quality of life due to the development of management skills with heart disease
Visits to the ED | 12 months
  Number of visits to the ED (Emergency Department) and/or hospitalizations during the follow-up period after the implantation of a defibrillator (ICD).
Mortality | 180 days
  Mortality rate at 180 days after the implantation of the ICD due to HF-related causes
Infection | 10 days
  Infection rate in the device pocket.

OTHER OUTCOMES:
Costs saving | 12 months
  How many costs are saved by the health system, the society, the patient, the caregiver and the hospital; thanks to Nursing therapeutics education.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Michela Gianino, Professor, Study Director — University of Turin, Italy; Sebastiano Marra, MD, Study Chair — University of Turin, Italy; Angela Durante, RN, Principal Investigator — Catholic University of Sacred Heart; Riccardo Sperlinga, MSC, Principal Investigator — Catholic Universit of Sacred Heart
Locations (2):
- Italy (2):
  - Cardiovascular Department, Rivoli Hospital, ASL TO3, Rivoli, Turin
  - Cardiovascular Department, Città della Salute e della Scienza, University Hospital, Turin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickey A, Barker M, McGee H, O'Boyle C. Measuring health-related quality of life in older patient populations: a review of current approaches. Pharmacoeconomics. 2005;23(10):971-93. doi: 10.2165/00019053-200523100-00002. PMID 16235972
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Pulignano G, Del Sindaco D, Minardi G, Tarantini L, Cioffi G, Bernardi L, Di Biagio D, Leonetti S, Giovannini E. Translation and validation of the Italian version of the European Heart Failure Self-care Behaviour Scale. J Cardiovasc Med (Hagerstown). 2010 Jul;11(7):493-8. doi: 10.2459/JCM.0b013e328335fbf5. PMID 20407384
- [Background] Stromberg A. Educating nurses and patients to manage heart failure. Eur J Cardiovasc Nurs. 2002 Feb;1(1):33-40. doi: 10.1016/S1474-5151(01)00011-1. PMID 14622865
- [Background] Aspromonte N, Di Tano G, Latini R, Masson S, Valle R, Emdin M. [Role of biomarkers for risk stratification in the tailored follow-up of heart failure patients]. G Ital Cardiol (Rome). 2010 May;11(5 Suppl 2):17S-23S. Italian. PMID 20873464
- [Result] MacIntyre K, Capewell S, Stewart S, Chalmers JW, Boyd J, Finlayson A, Redpath A, Pell JP, McMurray JJ. Evidence of improving prognosis in heart failure: trends in case fatality in 66 547 patients hospitalized between 1986 and 1995. Circulation. 2000 Sep 5;102(10):1126-31. doi: 10.1161/01.cir.102.10.1126. PMID 10973841
- [Result] Cocchieri A, Riegel B, D'Agostino F, Rocco G, Fida R, Alvaro R, Vellone E. Describing self-care in Italian adults with heart failure and identifying determinants of poor self-care. Eur J Cardiovasc Nurs. 2015 Apr;14(2):126-36. doi: 10.1177/1474515113518443. Epub 2013 Dec 23. PMID 24366984
- See also: Italian register for discharge — http://www.salute.gov.it/portale/documentazione/p6_2_8_3_1.jsp?lingua=italiano&id=16